CLINICAL TRIAL: NCT01285466
Title: A Phase Ib Multi-center, Open-label, 4-arm Dose-escalation Study of Oral BEZ235 and BKM120 in Combination With Weekly Paclitaxel in Patients With Advanced Solid Tumors and Weekly Paclitaxel/Trastuzumab in Patients With HER2+ Metastatic Breast Cancer
Brief Title: A Trial of Oral BEZ235 and BKM120 in Combination With Paclitaxel With or Without Trastuzumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235A2118; 2010-022331-11 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2017-02

CONDITIONS: Metastatic or Locally Advanced Solid Tumors
Keywords: Cancer; BEZ235; BKM120; paclitaxel; trastuzumab
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — dactolisib; Paclitaxel; NVP-BKM120; Trastuzumab

ARMS (4):
- BEZ235 + paclitaxel (Experimental)
  Interventions: Drug: BEZ235 + paclitaxel
- BKM120 + paclitaxel (Experimental)
  Interventions: Drug: BKM120 + paclitaxel
- BEZ235 + paclitaxel + trastuzumab (Experimental)
  Interventions: Drug: BEZ235 + paclitaxel + trastuzumab
- BKM120 + paclitaxel + trastuzumab (Experimental)
  Interventions: Drug: BKM120 + paclitaxel + trastuzumab

INTERVENTIONS:
Drug: BEZ235 + paclitaxel
  Arms: BEZ235 + paclitaxel
Drug: BKM120 + paclitaxel
  Arms: BKM120 + paclitaxel
Drug: BEZ235 + paclitaxel + trastuzumab
  Arms: BEZ235 + paclitaxel + trastuzumab
Drug: BKM120 + paclitaxel + trastuzumab
  Arms: BKM120 + paclitaxel + trastuzumab

SUMMARY:
The purpose of the trial is to determine the maximum tolerated dose (MTD) of BEZ235 and BKM120 in combination with weekly paclitaxel and weekly paclitaxel/trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with metastatic or locally advanced solid tumors, for whom weekly paclitaxel treatment is indicated (BEZ235-paclitaxel /BKM120-paclitaxel treatment)
* HER2+ metastatic or locally advanced breast cancer patients eligible for weekly paclitaxel and trastuzumab (BEZ235-paclitaxel-trastuzumab /BKM120-paclitaxel-trastuzumab treatment)
* Adult patients (≥ 18 years) (males, females)
* World Health Organization (WHO) performance status ≤ 2
* Adequate bone marrow function:
* Adequate hepatic and renal function:

Exclusion Criteria:

* Patients with primary central nervous system (CNS) tumor or CNS tumor involvement. However, patients with a metastatic CNS lesion may participate in this trial, if the patient is > 4 weeks from therapy (including radiation and/or surgery) completion, clinically stable with respect to the tumor at the time of study entry, and not receiving enzyme-inducing antiepileptic drugs or corticosteroid therapy or taper, as treatment of the brain metastases
* Patients who have received prior systemic anticancer therapy within the following time frames
* Cyclical chemotherapy: ≤ 3 weeks before study treatment (6 weeks for patients treated with nitrosoureas)
* Biological therapy: ≤ 4 weeks before study treatment, except treatment with trastuzumab (both parts of the trial)
* Investigational drug: ≤ 4 weeks before study treatment
* Patients who have undergone major surgery ≤ 4 weeks before study treatment
* Patients receiving chronic treatment with corticosteroids or other immunosuppressive agents
* Patients with uncontrolled, unmanageable, treatment-refractory diabetes mellitus
* Active or history of major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, history of suicide attempt or ideation, or homicide, as judged by the investigator and/or based on recent psychiatric assessment

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities during the first cycle of treatment. | First treatment cycle (4 weeks)

SECONDARY OUTCOMES:
Incidence of safety events during the whole treatment period (until progression of disease). | From start of treatment until disease progression
pharmacokinetics of BEZ235, BKM120 and paclitaxel given in combination, on Day 1, 8 and 22. | First treatment cycle (4 weeks)
Treatment efficacy (response to treatment according to RECIST criteria) | From start of treatment until disease progression
Impact of treatment on biomarkers of Pi3 Kinase pathway (analyses of skin biopsies, circulating markers) | From start of treatment until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Wilrijk
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Amsterdam, Netherlands
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
- Switzerland (2):
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Sankt Gallen

REFERENCES:
- See also: Results for CBEZ235A2118 can be found on the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14187